CLINICAL TRIAL: NCT04722003
Title: Mucosal Immune Responses Against Neisseria Gonorrhoeae Following Meningococcal Immunization in Healthy Young Adults
Brief Title: Mucosal Immunity Against Neisseria Gonorrhoeae After 4CMenB Vaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-0015
Record Dates: First submitted 2021-01-21; First posted 2021-01-25 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2020-12-11

CONDITIONS: Gonorrhoea
Keywords: 4CMenB; Gonorrhea; Meningococcal Group B Vaccine; Meningococcal Immunization; Mucosal Immune Response; Neisseria gonorrhoeae
MeSH Terms: conditions — Gonorrhea | interventions — 4CMenB vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 4CMenB (Experimental): Participants will receive two doses (0.5 mL each) of 4CMenB vaccine on Day 1 and Day 29. Each single dose of vaccine will be administered via intramuscular (IM) injection into the deltoid muscle of the preferred arm. N=40
  Interventions: Biological: Meningococcal Group B Vaccine
- Placebo (Placebo Comparator): Participants will receive two doses (0.5 mL each) of placebo injections (saline) on Day 1 and Day 29. Each single dose of placebo will be administered via intramuscular (IM) injection into the deltoid muscle of the preferred arm. N=10
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Meningococcal Group B Vaccine — A combination vaccine consisting of recombinant proteins Neisserial adhesin A (NadA), Neisserial Heparin Binding Antigen (NHBA), and factor H binding protein (fHbp), Outer Membrane Vesicles (OMV), aluminum hydroxide, sodium chloride, histidine, and sucrose.
  Arms: 4CMenB
Other: Placebo — 0.9% Sodium Chloride, USP injection.
  Arms: Placebo

SUMMARY:
This is a Phase 2 mechanistic clinical trial to assess the systemic and mucosal immunogenicity of the multicomponent meningococcal serogroup B vaccine (4CMenB or Bexsero (R)) (group 1, 40 subjects) against Neisseria gonorrhoeae, using a placebo vaccine (normal saline) as a comparator (group 2, 10 subjects). There will be approximately 50 participants, ages 18-49, both male and non-pregnant female subjects, enrolled at 1 site in the US. The goal will be to ensure adequate representation of subjects by sex in both treatment groups. The enrollment will be stratified by both sex and treatment arm. During enrollment of the "biopsy cohort" male and non-pregnant female subjects will be randomized 4:1 to either 4CMenB or placebo, up to a maximum of 10 male and 10 non-pregnant female subjects. Group 1 (approximate N=40) will receive two doses of 4CMenB on Day 1 and Day 29. Group 2 (approximate N=10) will receive two placebo injections on Day 1 and Day 29. Both groups will receive a single-dose prefilled syringe that is administered intramuscularly (0.5-mililiter each). The duration of each subject's participation is approximately 8 months, from recruitment through the last study visit, and the length of the study is estimated for 14 months. The primary objective is to characterize the rectal mucosal Immunoglobulin G IgG antibody response to Neisseria gonorrhoeae (GC) elicited by the 4CMenB vaccine as compared with the placebo vaccine (normal saline) in healthy adult subjects.

DETAILED DESCRIPTION:
This is a Phase 2 mechanistic clinical trial to assess the systemic and mucosal immunogenicity of the multicomponent meningococcal serogroup B vaccine (4CMenB or Bexsero (R)) (group 1, 40 subjects) against Neisseria gonorrhoeae, using a placebo vaccine (normal saline) as a comparator (group 2, 10 subjects). There will be approximately 50 participants, ages 18-49, both male and non-pregnant female subjects, enrolled at 1 site in the US. The goal will be to ensure adequate representation of subjects by sex in both treatment groups. The enrollment will be stratified by both sex and treatment arm. A subset of subjects in each treatment group (N=16 in Group 1, N=4 in Group 2) will undergo rectal mucosal biopsy at two time points (baseline and following the second vaccination) for assessment of tissue Neisseria gonorrhoeae (GC) specific cellular responses. During enrollment of the "biopsy cohort" male and non-pregnant female subjects will be randomized 4:1 to either 4CMenB or placebo, up to a maximum of 10 male and 10 non-pregnant female subjects. All subjects will undergo sampling of mucosal secretions for testing for antibodies against Neisseria gonorrhoeae (GC). Male subjects will undergo oropharyngeal and rectal mucosal sampling, and female subjects will undergo oropharyngeal, vaginal and rectal mucosal sampling. Group 1 (approximate N=40) will receive two doses of 4CMenB on Day 1 and Day 29. Group 2 (approximate N=10) will receive two placebo injections on Day 1 and Day 29. Both groups will receive a single-dose prefilled syringe that is administered intramuscularly (0.5-mililter each). The duration of each subject's participation is approximately 8 months, from recruitment through the last study visit, and the length of the study is estimated for 14 months. The primary objective is to characterize the rectal mucosal Immunoglobulin G (IgG) antibody response to Neisseria gonorrhoeae (GC) elicited by the 4CMenB vaccine as compared with the placebo vaccine (normal saline) in healthy adult subjects. The secondary objectives are: 1) To characterize the serum IgG antibody response to Neisseria gonorrhoeae (GC) elicited by the 4CMenB vaccine as compared with the placebo vaccine in healthy adult subjects, 2) To assess the safety and reactogenicity of 4CMenB in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Must be aged 18-49 years old (inclusive) at the time of vaccination.
2. Must be able to provide written informed consent.
3. Must have a body mass index (BMI) >/= 18.5 and < 35.0 kg/m2
4. Must be in good health based on physical examination, vital signs*, medical history, safety labs** (as applicable to the rectal biopsy and no biopsy cohorts) and the investigator's clinical judgment.

   *Vital signs must be within the normal ranges. If a subject has elevated systolic or diastolic blood pressure, subject may rest for 10 minutes in a quiet room and the blood pressure may be retaken.

   **Safety labs must be within the normal ranges and the normal ranges will be those used by the reference clinical lab.
5. For female subjects only: If a female participant is of childbearing potential*, she must use contraception** from 30 days before study product administration through the end of study participation.

   *A woman is considered of childbearing potential unless post-menopausal (defined as history of >/= 1 year of spontaneous amenorrhea), or permanently surgically sterilized (bilateral oophorectomy, salpingectomy, hysterectomy).

   **Acceptable methods of contraception include: abstinence or no sex with a male, monogamous relationship with a man who had a vasectomy at least 6 months before the 1st study vaccine, prescription oral contraceptives, intrauterine device (IUD), birth control implants or injections, contraceptive patch, vaginal ring, condoms and diaphragms/cervical cap with spermicide ("double barrier" method).
6. Must be available and willing to participate for the duration of this trial.
7. Willing to provide mucosal samples: vaginal secretions for women and oropharyngeal and rectal secretions for men and women.
8. For the rectal biopsy cohort only, willing to provide rectal biopsies.

Exclusion Criteria:

1. Has ever been diagnosed with meningococcal infection or gonococcal infection at any anatomic site.
2. Has ever received any serogroup B meningococcal vaccine.
3. Any positive test result for STI (including Neisseria gonorrhoeae (GC) Chlamydia trachomatis (CT), Rapid Plasma Reagin (RPR) and Human Immunodeficiency Virus (HIV)) at screening*.

   *Female subjects will also be tested for Trichomonas at screening.
4. Any history of Chlamydia trachomatis or syphilis infection at any body site in the preceding 12 months
5. Has known allergy or history of anaphylaxis or other serious adverse reaction to a vaccine or vaccine products.
6. Has severe allergy or anaphylaxis to latex.
7. Has an acute illness or temperature >/= 38.0 degrees Celsius on Day 1*.

   *Subjects with fever or acute illness on the day of vaccination may be re-assessed and enrolled if healthy or only minor residual symptoms remain within 3 days.
8. Has a history of a bleeding disorder, or is taking chronic anti-coagulant (e.g. warfarin, direct thrombin inhibitors, heparin products, etc.), anti-platelet, or non-steroidal anti-inflammatory drugs (NSAID) therapy.
9. Has history of autoimmune disease, or clinically significant cardiac, pulmonary, gastrointestinal, hepatic, rheumatologic, or renal disease by history or physical examination.
10. Has history of active malignancy other than squamous cell or basal cell skin cancer, unless there has been surgical excision that is considered to have achieved cure*.

    *Subjects with a history of skin cancer must not be vaccinated at the previous tumor site.
11. Has known or suspected congenital or acquired immunodeficiency, or recent history or current use of immunosuppressive therapy*.

    *Anti-cancer chemotherapy or radiation therapy within the preceding 3 years, or long-term (>/= 2 weeks within the previous 3 months) systemic corticosteroid therapy (at a dosage of >/= 0.5 mg/kg/day). Intranasal or topical prednisone (or equivalent) are allowed.
12. Is post-organ and/or stem cell transplant, whether or not on chronic immunosuppressive therapy.
13. Had major surgery (per the investigator's judgment) within 4 weeks before study entry or planned major surgery during this trial.
14. Has history of diabetes* mellitus type 1 or type 2, including cases controlled with diet alone*.

    *History of isolated gestational diabetes is not an exclusion criterion.
15. Received live attenuated vaccines from 30 days before first vaccination until 30 days after second vaccination.
16. Received killed or inactivated vaccines* from 14 days before first vaccination until 14 days after second vaccination.

    *For inactivated influenza vaccine, from 7 days before either vaccination until 7 days after either vaccination.
17. Received mRNA, viral vector, or any other technology platform Corona Virus Disease-19 (COVID-19) vaccine within 14 days prior to first dose of the study product.*

    *COVID-19 vaccination should take priority over administration of the study product.
18. Received experimental therapeutic agents within 12 months before first vaccination or plans to receive any experimental therapeutic agents during this trial except for Emergency Use Authorization (EUA) COVID-19 therapy.*

    *Only exclusionary if, in the opinion of the investigator, they would interfere with safety or endpoint assessment.
19. Is currently participating or plans to participate in another clinical study which would involve receipt of an investigational product or undergoing a procedure*.

    *Only exclusionary if, in the opinion of the investigator, they would interfere with safety or endpoint assessment.
20. Received blood products or immunoglobulin in the 3 months before study entry or planned use during this trial.
21. Has major psychiatric illness in the past 12 months that in the opinion of the investigator would preclude participation.
22. Has current alcohol use or current or past abuse of recreational or narcotic drugs by history as judged by the investigator to potentially interfere with study adherence.
23. In the opinion of the investigator cannot communicate reliably, is unlikely to adhere to the requirements of this trial, or has any condition which would limit the ability to complete this trial.
24. Is pregnant or breast feeding.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hope Clinic of Emory University, Decatur, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were males and non-pregnant females, 18 to 49 years of age, inclusive, who were in good health and meet all eligibility criteria.
Groups:
- 4CMenB: Participants will receive two doses (0.5 mL each) of 4CMenB vaccine on Day 1 and Day 29. Each single dose of vaccine will be administered via intramuscular (IM) injection into the deltoid muscle of the preferred arm.
  Meningococcal Group B Vaccine: A combination vaccine consisting of recombinant proteins Neisserial adhesin A (NadA), Neisserial Heparin Binding Antigen (NHBA), and factor H binding protein (fHbp), Outer Membrane Vesicles (OMV), aluminum hydroxide, sodium chloride, histidine, and sucrose.
- Placebo: Participants will receive two doses (0.5 mL each) of placebo injections (saline) on Day 1 and Day 29. Each single dose of placebo will be administered via intramuscular (IM) injection into the deltoid muscle of the preferred arm.
  Placebo: 0.9% Sodium Chloride, USP injection.
Period: Overall Study
Arm/Group | 4CMenB | Placebo
Started | 41 | 11
Completed | 38 | 11
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 4CMenB | Placebo | Total
Number analyzed (Participants) | 41 | 11 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (7.5) | 29.8 (8.1) | 31.1 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 6 | 27
  Male | 20 | 5 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 36 | 9 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 10 | 2 | 12
  White | 21 | 7 | 28
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Rectal Mucosal IgG Concentrations (Geometric Mean Titers [GMT]) Against N. Gonorrhoeae Outer Membrane Vesicle (OMV) Antigen Ng1291
Description: Rectal mucosal IgG concentrations (geometric mean titers, GMT) against GC OMV antigen Ng1291 by ELISA at Day 1, 29, 43, 57, and 181 in each treatment group
Time Frame: Day 1 through Day 181
Population: Immunogenicity Population: For the primary outcome analysis, the immunogenicity population at a specified follow-up visit will include all eligible participants who have received all doses of study product prior to that visit and have immunogenicity data available for that visit. Which includes all participants who received at least one dose of study vaccine and contributed at least one sample for immunogenicity testing for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 4CMenB | Placebo
Number analyzed (Participants) | 40 | 11
titer
  Day 1: number analyzed (Participants) | 12 | 8
  Day 1 | 0.07 [0.027 to 0.182] | 0.072 [0.025 to 0.213]
  Day 29: number analyzed (Participants) | 16 | 7
  Day 29 | 0.089 [0.041 to 0.192] | 0.097 [0.056 to 0.167]
  Day 43: number analyzed (Participants) | 23 | 4
  Day 43 | 0.078 [0.046 to 0.133] | 0.047 [0.024 to 0.09]
  Day 57: number analyzed (Participants) | 24 | 4
  Day 57 | 0.135 [0.095 to 0.192] | 0.062 [0.028 to 0.137]
  Day 181: number analyzed (Participants) | 23 | 7
  Day 181 | 0.182 [0.123 to 0.268] | 0.055 [0.03 to 0.1]

2. Primary Outcome: Rectal Mucosal IgG Concentrations (Geometric Mean Titers [GMT]) Against N. Gonorrhoeae Outer Membrane Vesicle (OMV) Antigen CNG20
Description: Rectal mucosal IgG concentrations (geometric mean titers, GMT) against GC OMV antigen CNG20 by ELISA at Day 1, 29, 43, 57, and 181 in each treatment group
Time Frame: Day 1 through day 181
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 4CMenB | Placebo
Number analyzed (Participants) | 40 | 11
titer
  Day 1: number analyzed (Participants) | 19 | 9
  Day 1 | 0.125 [0.063 to 0.25] | 0.156 [0.07 to 0.345]
  Day 29: number analyzed (Participants) | 23 | 7
  Day 29 | 0.165 [0.086 to 0.318] | 0.104 [0.042 to 0.255]
  Day 43: number analyzed (Participants) | 27 | 5
  Day 43 | 0.136 [0.084 to 0.221] | 0.087 [0.039 to 0.195]
  Day 57: number analyzed (Participants) | 29 | 8
  Day 57 | 0.181 [0.113 to 0.29] | 0.048 [0.025 to 0.093]
  Day 181: number analyzed (Participants) | 27 | 8
  Day 181 | 0.207 [0.128 to 0.333] | 0.066 [0.037 to 0.119]

3. Secondary Outcome: Serum IgG Concentrations (Geometric Mean Titers [GMT]) Against N. Gonorrhoeae Outer Membrane Vesicle (OMV) Antigen Ng1291
Description: Serum IgG concentrations (geometric mean titers, GMT) against GC OMV antigen Ng1291 at Day 1, 29, 43, 57, and 181 in each treatment group
Time Frame: Day 1 through Day 181
Population: Immunogenicity Population: The immunogenicity population at a specified follow-up visit will include all eligible participants who have received all doses of study product prior to that visit and have immunogenicity data available for that visit. Which includes all participants who received at least one dose of study vaccine and contributed at least one sample for immunogenicity testing for which valid results were reported.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 4CMenB | Placebo
Number analyzed (Participants) | 40 | 11
titer
  Day 1 | 75.233 [54.898 to 103.101] | 144.85 [99.992 to 209.832]
  Day 29: number analyzed (Participants) | 40 | 10
  Day 29 | 227.844 [176.002 to 294.956] | 154.356 [96.714 to 246.352]
  Day 43: number analyzed (Participants) | 40 | 10
  Day 43 | 324.931 [267.057 to 395.347] | 143.878 [94.851 to 218.245]
  Day 57: number analyzed (Participants) | 39 | 10
  Day 57 | 301.169 [246.083 to 368.585] | 156.602 [108.694 to 225.626]
  Day 181: number analyzed (Participants) | 38 | 11
  Day 181 | 163.493 [131.056 to 203.958] | 143 [92.976 to 219.938]

4. Secondary Outcome: Serum IgG Concentrations (Geometric Mean Titers [GMT]) Against N. Gonorrhoeae Outer Membrane Vesicle (OMV) Antigen CNG20
Description: Serum IgG concentrations (geometric mean titers, GMT) against GC OMV antigen CNG20 at Day 1, 29, 43, 57, and 181 in each treatment group
Time Frame: Day 1 through day 181
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 4CMenB | Placebo
Number analyzed (Participants) | 40 | 11
titer
  Day 1 | 50.09 [34.906 to 71.877] | 90.931 [58.09 to 142.338]
  Day 29: number analyzed (Participants) | 40 | 10
  Day 29 | 181.509 [136.805 to 240.82] | 89.334 [56.738 to 140.658]
  Day 43: number analyzed (Participants) | 40 | 10
  Day 43 | 292.209 [238.827 to 357.524] | 86.342 [53.586 to 139.122]
  Day 57: number analyzed (Participants) | 39 | 10
  Day 57 | 262.937 [215.848 to 320.298] | 90.205 [55.521 to 146.556]
  Day 181: number analyzed (Participants) | 38 | 11
  Day 181 | 136.722 [108.9 to 171.653] | 100.148 [61.631 to 162.735]

5. Secondary Outcome: The Reactogenicity of 4CMenB in Healthy Adult Participants
Description: Frequency and severity of any adverse events (AE) related to 4CMenB immunization
Time Frame: Day 1 through Day 181
Population: The safety analysis population includes all participants who received at least one dose of study treatment. For analyses using the safety population, participants will be grouped by study treatment received
Measure: Count of Participants; unit: Participants
Arm/Group | 4CMenB | Placebo
Number analyzed (Participants) | 41 | 11
Participants
  Any Symptom: number analyzed (Participants) | 41 | 6
  Any Symptom: Mild | 12 | 5
  Any Symptom: Moderate | 24 | 1
  Any Symptom: Severe | 5 | 0
  Any Systemic Symptom: number analyzed (Participants) | 39 | 5
  Any Systemic Symptom: Mild | 24 | 4
  Any Systemic Symptom: Moderate | 12 | 1
  Any Systemic Symptom: Severe | 3 | 0
  Arthralgia: number analyzed (Participants) | 8 | 0
  Arthralgia: Mild | 5 | 0
  Arthralgia: Moderate | 3 | 0
  Arthralgia: Severe | 0 | 0
  Fatigue: number analyzed (Participants) | 25 | 1
  Fatigue: Mild | 17 | 1
  Fatigue: Moderate | 6 | 0
  Fatigue: Severe | 2 | 0
  Headache: number analyzed (Participants) | 19 | 5
  Headache: Mild | 16 | 4
  Headache: Moderate | 3 | 1
  Headache: Severe | 0 | 0
  Malaise: number analyzed (Participants) | 20 | 0
  Malaise: Mild | 15 | 0
  Malaise: Moderate | 3 | 0
  Malaise: Severe | 2 | 0
  Myalgia: number analyzed (Participants) | 26 | 0
  Myalgia: Mild | 21 | 0
  Myalgia: Moderate | 4 | 0
  Myalgia: Severe | 1 | 0
  Nausea: number analyzed (Participants) | 6 | 0
  Nausea: Mild | 4 | 0
  Nausea: Moderate | 1 | 0
  Nausea: Severe | 1 | 0
  Pyrexia: number analyzed (Participants) | 13 | 0
  Pyrexia: Mild | 7 | 0
  Pyrexia: Moderate | 4 | 0
  Pyrexia: Severe | 2 | 0
  Any Local Symptom: number analyzed (Participants) | 40 | 2
  Any Local Symptom: Mild | 12 | 2
  Any Local Symptom: Moderate | 24 | 0
  Any Local Symptom: Severe | 4 | 0
  Administration Site Bruise: number analyzed (Participants) | 3 | 1
  Administration Site Bruise: Mild | 3 | 1
  Administration Site Bruise: Moderate | 0 | 0
  Administration Site Bruise: Severe | 0 | 0
  Administration Site Erythema: number analyzed (Participants) | 8 | 0
  Administration Site Erythema: Mild | 6 | 0
  Administration Site Erythema: Moderate | 2 | 0
  Administration Site Erythema: Severe | 0 | 0
  Administration Site Induration: number analyzed (Participants) | 10 | 0
  Administration Site Induration: Mild | 8 | 0
  Administration Site Induration: Moderate | 1 | 0
  Administration Site Induration: Severe | 1 | 0
  Administration Site Pain: number analyzed (Participants) | 38 | 0
  Administration Site Pain: Mild | 22 | 0
  Administration Site Pain: Moderate | 15 | 0
  Administration Site Pain: Severe | 1 | 0
  Administration Site Pruritus: number analyzed (Participants) | 3 | 0
  Administration Site Pruritus: Mild | 3 | 0
  Administration Site Pruritus: Moderate | 0 | 0
  Administration Site Pruritus: Severe | 0 | 0
  Administration Site Tenderness: number analyzed (Participants) | 40 | 1
  Administration Site Tenderness: Mild | 16 | 1
  Administration Site Tenderness: Moderate | 21 | 0
  Administration Site Tenderness: Severe | 3 | 0

6. Secondary Outcome: Frequency of Serious Adverse Events (SAE)
Description: Frequency of SAEs through the end of the study.
Time Frame: Day 1 through Day 181
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | 4CMenB | Placebo
Number analyzed (Participants) | 41 | 11
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited injection site and systemic reactogenicity events were documented and reported from Day 1 through Day 8 and Day 29 through Day 36. Unsolicited AEs were collected and assessed through the end of the protocol-defined follow up period (181 days post first vaccination)
Arm/Group | 4CMenB | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/11
Other Adverse Events (participants affected / at risk) | 41/41 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 4CMenB (N=41) | Placebo (N=11)
Administration site bruise (General disorders) | 3 (3) | 1 (1)
Administration site erythema (General disorders) | 8 (9) | 0 (0)
Administration site induration (General disorders) | 10 (14) | 0 (0)
Administration site pain (General disorders) | 38 (68) | 0 (0)
Administration site pruritus (General disorders) | 3 (4) | 0 (0)
Administration site tenderness (General disorders) | 40 (77) | 1 (2)
Fatigue (General disorders) | 25 (38) | 1 (2)
Malaise (General disorders) | 20 (24) | 0 (0)
Pyrexia (General disorders) | 13 (16) | 0 (0)
Arthraliga (Musculoskeletal and connective tissue disorders) | 8 (12) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 26 (36) | 0 (0)
Headache (Nervous system disorders) | 19 (25) | 5 (6)
Nausea (Gastrointestinal disorders) | 6 (7) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abnormal uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2023-08-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT04722003/Prot_001.pdf
  • Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/03/NCT04722003/SAP_002.pdf
  • Informed Consent Form (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/03/NCT04722003/ICF_000.pdf